CLINICAL TRIAL: NCT00142714
Title: Effects of SCI on Female Sexual Response
Brief Title: Effects of Spinal Cord Injury on Female Sexual Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 5R01HD030149-09 (NIH)
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2006-10-16 (Estimated); Status verified 2006-10

CONDITIONS: Female Sexual Dysfunction; Multiple Sclerosis; Spinal Cord Injury
Keywords: sexual response; sexual dysfunction in females; spinal cord injury
MeSH Terms: conditions — Multiple Sclerosis; Spinal Cord Injuries

INTERVENTIONS:
Procedure: Sympathetic manipulation on sexual arousal in women

SUMMARY:
The long term aims of this project are to 1) Understand the effect of varying degrees and levels of SCI and dysfunction(SCI/D)on females sexual response: 2) Identify the specific neuronal pathways involved in female sexual responses; and 3) Develop and evaluate new assessment and treatment methods for neurogenic sexual dysfunction in women.

ELIGIBILITY:
Inclusion Criteria:

* MS or SCI
* Normal menstrual periods
* Normal hand function
* Have ability to feel sensation from lower abdomen to upper thigh region.

Exclusion Criteria:

* Pregnant
* Menopausal

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70
Dates: Start 2003-08; Study Completion 2005-06

PRIMARY OUTCOMES:
Our central hypothesis are:
1) In females the SNS regulates psychogenic genital vasocongestion 2) In females the orgasmic reflex requires the presence of an intact sacral spinal cord, 3) In females a pattern generator is responsible for the orgasmic reflex.

CONTACTS AND LOCATIONS:
Overall Officials: Marca Sipski, MD, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- The University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Alexander M, Bashir K, Alexander C, Marson L, Rosen R. Randomized Trial of Clitoral Vacuum Suction Versus Vibratory Stimulation in Neurogenic Female Orgasmic Dysfunction. Arch Phys Med Rehabil. 2018 Feb;99(2):299-305. doi: 10.1016/j.apmr.2017.09.001. Epub 2017 Sep 9. PMID 28899827